CLINICAL TRIAL: NCT06126198
Title: 1 Hz RTMS Feasibility Study on Adolescent Treatment Resistant Major Depression
Brief Title: RTMS Feasibility Study on Adolescent Depression Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: Uppsala University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Teen-TMS_UU2023
Record Dates: First submitted 2023-11-03; First posted 2023-11-13 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Major Depressive Disorder; Unipolar Depression; Bipolar Depression
Keywords: repetitive transcranial magnetic stimulation
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder; Bipolar Disorder | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Open label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Active treatment (Experimental): Active treatment with Repetitive Transcranial Magnetic Stimulation (rTMS) according to clinical protocol.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation (rTMS) — rTMS induces local electrical currents in the stimulated neurons and has been shown to induce long-term inhibition or excitation of groups of neurons in treated cortical areas

SUMMARY:
This is an open-label study, in which all participants receives an active treatment with repetitive transcranial magnetic stimulation (rTMS) according to clinical protocol. The aim with this pilotstudy is to investigate the feasibility to perform a trial of low-frequency rTMS on treatment-resistant depression in adolescents. The study includes adolescents 13-19 years old, with average to severe depression.

DETAILED DESCRIPTION:
The intervention follows the identical clinical procedure used for adults. Initially, the resting motor threshold will be determined by stimulation over the motor cortex, by finding the minimal intensity that produces a motor response in the corresponding distal wrist muscles. The rTMS will be delivered with a powerMAG research ppTMS stimulator (Mag & More), and a figure-of -eight coil, PMD70-pCool (Mag & More). The intervention is within the intended use of this CE-marked medical device. The research participants will receive 1Hz rTMS with daily sessions on 20-30 consecutive week days. The magnetic pulses will be applied at 120% of the resting motor threshold with a figure-of-eight coil at a 45 degree angle towards the midline. The 1Hz rTMS protocol is applied 6 trains of 1-min duration separated by 30-sec inter-train "off" periods over the right DLPFC (F4 site 5 according to the10-20 system). The total duration of one 1 Hz rTMS session is 8 min 30 s.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent from parents and legal guardian
* Age 13-19 years
* Diagnosis of uni- or bipolar depression verified through a Mini International Neuropsychiatric Interview for children and adolescents (MINI-KID)
* Treatment with at least two SSRIs at an adequate dose for at least 8 weeks

Exclusion Criteria:

* Epilepsy or medical history of seizures
* Conductive ferromagnetic or other magnetic sensitive metals implanted in the head or within 30 cm of the treatment coil
* Implanted device that is activated or controlled in any way by physiological signals
* Implanted medication pumps
* Intracardiac lines (even if removed)
* Active substance use disorder
* Treatment with any medication that could lower the threshold for seizures
* Usage of benzodiazepines both as prescribed drug and illegal use
* Any condition that seriously increases the risk of non-compliance or loss of follow-up

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Inclusion rate - | two years
  Participant inclusion during the course of the study
Attrition rate | two years
  Participant drop-off during the course of the study

SECONDARY OUTCOMES:
CGAS (Children's Global Assessment Scale) score | 4 weeks, 6 weeks
  Children's Global Assessment Scale, score 1-100, where a high score indicates high functioning.
MADRS (Montgomery and Asberg Depression Rating Scale) score | at Baseline, 4 weeks, 6 weeks
  Montgomery and Asberg Depression Rating Scale, score 0-60, where a high score indicates symtoms of depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Uppsala University, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No